CLINICAL TRIAL: NCT06648655
Title: A Phase 2, Randomized, Investigator and Participant bLInded, placeBo-controllEd, paRallel-group Study to Investigate the sAfety, Tolerability, and Preliminary Efficacy of TMP-301 TrEatment in Adult Patients With Alcohol Use Disorder (AUD)
Brief Title: A Study to Investigate the Safety and Efficacy of TMP-301 Compared to Placebo in Adult Patients With Alcohol Use Disorder
Acronym: LIBERATE-A
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tempero Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMP-301-AUD-201
Record Dates: First submitted 2024-10-10; First posted 2024-10-18 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: AUD; Substance Use Disorders; SUD
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TMP-301 (Experimental): Daily (QD) x 14 weeks.
  Interventions: Drug: TMP-301
- Placebo (Placebo Comparator): Daily (QD) x 14 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TMP-301 — Daily (QD) x 14 weeks.
  Arms: TMP-301
Drug: Placebo — Daily (QD) x 14 weeks.
  Arms: Placebo

SUMMARY:
TMP-301 has been shown in preclinical models to reduce consumption of alcohol and other addictive substances. It has been tested in healthy subjects and has been found to be safe and tolerated at doses predicted to be efficacious in alcohol use disorder. This study is being conducted to evaluate the safety, tolerability and efficacy of TMP-301 in patients with alcohol use disorder.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability and effect on alcohol use (number of heavy drinking days) of TMP-301 compared to placebo in patients with alcohol use disorder. This is a placebo-controlled, parallel-group, multicenter clinical study in moderate to severe alcohol use disorder with ≥8 heavy drinking days over the prior 4 weeks at screening. Study participants and investigators will be blinded to study intervention. The study duration will be up to 19 weeks, with a treatment duration of up to 14 weeks. The visit frequency will be weekly.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated Informed Consent Form (ICF) with a stated willingness to comply with all study procedures and availability for the duration of the study. A breathalyzer test must be <0.05% at the time of ICF signing. Participants who have a blood alcohol content between 0.02 and 0.04% inclusive at Screening will be assessed for competency to consent using the UBACC scale. Participants must have a passing score of ≥ 15 during the Screening period to consent and be eligible for randomization.
2. Adult female or male, 18 to 65 years of age inclusive, at the time of screening.
3. Alcohol use disorder, moderate or severe by DSM-5 diagnostic criteria (i.e., ≥4 out of 11 symptoms present using the SCID-5-CT diagnostic interview) at screening for the previous 12 months.
4. At least 8 heavy drinking days over the previous 4 weeks (by Timeline Follow Back) at screening.

   * Heavy Drinking Days (HDD): ≥4 drinks/day for females, ≥5 drinks/ day for males.
   * A standard drink is defined as 12 ounces (350 ml) of 5% beer, 5 ounces (150 ml) of 12% wine, or 1.5 ounces (44 ml) of 80-proof (40%) distilled spirits.
5. Seeking treatment for AUD, with a desire to reduce or cease alcohol use at screening.
6. Breathalyzer <0.05% at baseline..
7. BMI of ≥18.0 to ≤40.0 kg/m2 at screening.
8. No clinically significant findings (in the investigator's opinion) on physical exam, ECG, vital signs, or clinical laboratory tests at screening. The following criteria must be met:

   * Systolic Blood Pressure (SBP) 90-140 mmHg, and Diastolic Blood Pressure (DBP) 50-90 mmHg, inclusive (average of three readings) at screening and baseline.
   * Alanine transaminase (ALT) and Aspartate transferase (AST) < 3x upper limit of normal, and total bilirubin < upper limit of normal (isolated elevated total bilirubin is allowed if Gilbert's syndrome is the suspected etiology)..
   * Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73 m2
   * Negative urine drug screen for cocaine or stimulants at screening and baseline
9. Able to communicate well and understand written instructions.
10. Agree to practice highly effective birth control starting at screening and continuing for 30 days (females) or 90 days (males) after study treatment ends.

    1. For females any of the following (no donation of eggs/ova is allowed):

       * Abstinence from heterosexual intercourse.
       * Postmenopausal: absence of menses ≥ 12 months (without an alternative medical condition) and Follicle-Stimulating Hormone (FSH) ≥ 40 mIU/mL at screening.
       * Surgically sterile: bilateral oophorectomy, salpingectomy, tubal ligation, or hysterectomy ≥180 days prior to screening.
       * Contraceptive implant or intrauterine device.
    2. For males any of the following (no donation of sperm is allowed):

       * Abstinence from heterosexual intercourse.
       * Male condom with spermicide or male condom with vaginal spermicide (gel, foam, or suppository).
       * Surgically sterile: post vasectomy or bilateral orchiectomy

Exclusion Criteria:

1. History of hypersensitivity to TMP-301 or other mGluR5 antagonists.
2. Evidence of suicidal risk as assessed by the Columbia-Suicide Severity Rating Scale at screening or baseline as follows:

   * Suicidal Ideation Section: "Yes" on item 4 or 5 if within 6 months of screening or between screening and baseline.
   * Suicidal Behavior Section: "Yes" on any item (except non-suicidal self-injurious behavior) if within 2 years of screening or between screening and baseline.
3. Significant risk of acute alcohol withdrawal syndrome (either of the following):

   * Any history of Delirium Tremens or seizures from alcohol withdrawal.
   * Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) score >7 at screening or baseline.
4. Any history of seizures, except febrile seizures as a child.
5. Other (non-alcohol) substance use disorders (by DSM-5) as follows:

   * Any cocaine or stimulant use disorder
   * Moderate or severe use disorder of all other substances (mild allowed).
6. Use of the following within the last 90 days or ≥ 5 times the half-life prior to randomization:

   * Pharmacotherapy for any substance use disorder (e.g.: disulfiram, acamprosate, modafinil, topiramate, or baclofen).
   * Use of prescribed methylphenidate or other stimulant.
   * Use of any Glucagon-like peptide 1 (GLP-1) agonist for any indication.
7. Past or current history of any mental, behavioral, or neurodevelopmental disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) or significant risk of developing a psychosis (assessed by PRIME screen) or a personal history of psychotic symptoms (hallucinations or delusions) with or without a formal psychiatric diagnosis.

   * Individuals with AUD or mild other substance use disorder (except for cocaine or stimulants) may participate.
   * Individuals who meet criteria for a current major depressive episode are excluded.
8. Requires treatment with any psychoactive medications, including any anti-seizure medications (except medications used for short-term treatment of insomnia).

   - Antidepressant medications are allowed if the patients have been on an adequate and stable dose for at least 3 months prior to study treatment dosing with the exception of CYP1A2 substrates or CYP3A4 inhibitors as detailed in Exclusion 19.
9. Having had initiation of, or change in intensity of, psychotherapy or other non-drug therapies within 6 weeks prior to enrollment or unwillingness to maintain current psychotherapeutic and non-drug therapy levels from screening through the or at any time during the acute treatment phase of the study.
10. Use of other investigational drugs or devices at the time of screening, or within 5 half-lives of randomization, or within 30 days, whichever is longer or has been part of any clinical study within 30 days of randomization.
11. Pregnant or nursing (lactating) females.
12. Recent history or active clinically significant manifestations of metabolic, hepatic, renal (including porphyria), hematological, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, dermatological, urogenital, neurological, ophthalmic, or ears, nose, and throat (ENT) disorders, or any other acute or chronic condition or medication use that, in the Investigator's opinion, would limit the subject's ability to complete or participate in this clinical study.
13. Concomitant use of agents known to prolong the QT interval unless these can be permanently discontinued for the duration of study.
14. History or current diagnosis of ECG abnormalities at screening indicating significant risk of safety for subjects participating in the study such as:

    * Concomitant clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia, and clinically significant second- or third-degree Atrioventricular (AV) block without a pacemaker.
    * History of familial long QT syndrome or known family history of Torsades de Pointes.
    * QTcF > 450 msec (males); QTcF > 460 msec (females).
    * Note: sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are not exclusionary.
15. Patients with history of chronic hypertension, unless well controlled by taking antihypertensive treatment at a stable dose for ≥3 months
16. History or presence of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there was evidence of local recurrence or metastases.
17. Detectable hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV) antibody at screening.

    - Participants in remission for HCV or HIV, as demonstrated by a sustained virological response (undetectable viral load) may be enrolled in the study.
18. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
19. Need/plan to take or substrates of cytochrome P450 (CYP)1A2 or inhibitors of CYP3A4. (Note: CYP1A2 inhibitors are permitted, as they are not expected to increase TMP-301 exposures above what was shown to be safe and generally well-tolerated in study TMP-301- HNV-101.).

    * CYP1A2 Substrates: (Exposure could increase when taken with TMP-301):
    * alosetron, duloxetine, melatonin, ramelteon, tasimelteon, tizanidine, pimozide, agomelatine, tacrine, clozapine, pirfenidone, theophylline, tacrine, ropivacaine
    * CYP3A4 Inhibitors: Could increase TMP-301 exposure at steady- state
    * grapefruit juice, Seville orange-containing food (e.g. bitter orange marmalade) or drink (e.g. bitter orange liqueurs including Curaçao and Grand Marnier)
    * ketoconazole, diltiazem, verapamil, clarithromycin, itraconazole, erythromycin, fluconazole, ceritinib, cobicistat, idelalisib, indinavir. ritonavir, nefazodone, lopinavir, aprepitant, ciprofloxacin, conivaptan, crizotinib, dronedarone, imatinib
20. Patient cannot:

    * Anticipate any significant problems with transportation arrangements or available time to travel to the study site and have any plans to move within the next months to a location which would make continued participation in the study' impractical.
    * Be involved in any unresolved legal problems that could jeopardize continuation or completion of the study.
    * Have any pending charges for violent crime (not including Driving Under the Influence (DUI) offenses).
    * Have any court case with a pending decision that could prohibit participation or compliance in the study.
21. Living situation precludes an ability to adhere to study visits in the opinion of the investigator.
22. Has been previously treated in this study or randomized or treated in any other study employing TMP-301 (i.e., subject may not have received study drug and then reenrolled).
23. Any condition not identified in the protocol that in the opinion of the investigator would confound the evaluation and interpretation of the study data or may put the subject at risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of TMP-301 in patients with alcohol use disorder | Baseline to Week 16
  To evaluate the safety and tolerability of TMP-301 in patients with alcohol use disorder by the incidence and severity of Adverse Events
To evaluate the efficacy of TMP-301 in patients with alcohol use disorder as assessed by the Timeline to Followback measurement | Baseline to Week 14
  The Timeline Followback (TLFB) instrument/measurement is used as a clinical tool to obtain quantitative estimates of alcohol use.

SECONDARY OUTCOMES:
To evaluate the effect of TMP-301 on the number of days that alcohol is consumed | Baseline to Week 14
To evaluate the effect of TMP-301 on abstinence from alcohol use | Baseline to Week 14
  Subjects will be asked if they have consumed alcohol.
To evaluate the effect of TMP-301 on number of no heavy drinking days | Baseline to Week 14
  Subjects will be asked about heavy drinking days, defined as ≥4 drinks/day for females, ≥5 drinks/day for males.
To evaluate the effect of TMP-301 on improvement in world health organization risk score | Baseline to Week 14
To evaluate plasma TMP-301 concentrations in patients with alcohol use disorder | Baseline to Week 14
  To evaluate Ctrough of TMP-301 concentrations in patients with alcohol use disorder
To evaluate plasma TMP-301 concentrations in patients with alcohol use disorder | Baseline to Week 14
  To evaluate C2hr of TMP-301 concentrations in patients with alcohol use disorder

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Headlands Research, Scottsdale, Arizona
  - Yale School of Medicine, New Haven, Connecticut
  - Research Centers of America, LLC, Hollywood, Florida
  - CNS Healthcare- Jacksonville South, Jacksonville, Florida
  - Segal Trials - West Broward Outpatient Site, Lauderhill, Florida
  - CNS Healthcare, Orlando, Florida
  - CenExcel iResearch, Decatur, Georgia
  - CenExcel iResearch, Savannah, Georgia
  - DelRicht Research - Murphy Clinic, Mandeville, Louisiana
  - IMA Clinical Research, Albuquerque, New Mexico
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Medical University of South Carolina, Institute of Psychiatry, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia: Center for Leading Edge Addiction Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No